CLINICAL TRIAL: NCT01915472
Title: A Phase II Study of IMMU 130 (hMN-14-SN38 Antibody Drug Conjugate) in Patients With Metastatic Colorectal Cancer
Brief Title: A Phase II Study of IMMU 130 in Patients With Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMU 130-03
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Colorectal Cancer; Rectal Cancer; previously treated
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Immunoconjugates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMMU 130 (Experimental)
  Interventions: Drug: IMMU 130

INTERVENTIONS:
Drug: IMMU 130 — This is a Phase II, open-label study of IMMU-130 administered every 14 days for a period of 24 weeks to patients with metastatic colorectal cancer who have been previously treated with at least one prior irinotecan-containing regimen.
  Other Names: hMN14-SN38; Labetuzumab-SN38; antibody-drug conjugate

SUMMARY:
This is a Phase II trial to study the safety and efficacy of IMMU-130. IMMU-130 is composed of a drug attached to an antibody. The drug is the active ingredient in irinotecan which is a common chemotherapy drug used for colorectal cancer. Antibodies are proteins normally made by the immune system. They bind to substances that don't belong in the body to prevent harm to the body. The antibody in this study was designed to bind to a marker located on colorectal cancer tumors. The antibody was originally made from mouse proteins, but was changed in the laboratory to be more like human antibodies. This study will investigate how IMMU-130 acts for the treatment of colorectal cancer. The study is mainly being done to see if IMMU-130 is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥ 18 years of age, able to understand and give written informed consent
* Histologically or cytologically confirmed colorectal adenocarcinoma
* Stage IV (metastatic) disease
* Previously treated with at least one prior irinotecan-containing regimen for colorectal cancer
* Adequate performance status (ECOG 0 or 1) (Appendix 1)
* Expected survival ≥ 6 months
* CEA plasma levels > 5 ng/mL
* Measurable disease by CT or MRI, but with no single lesion measuring more than 10.0 cm
* At least 4 weeks beyond treatment (chemotherapy, immunotherapy and/or radiation therapy) or major surgery and recovered from all acute toxicities
* Adequate hematology without ongoing transfusional support (hemoglobin > 8 g/dL, ANC ≥ 1,500 per mm3, platelets > 100,000 per mm3)
* Adequate renal and hepatic function (creatinine ≤ 1.5 x IULN, bilirubin within normal limits, AST and ALT ≤ 3.0 x IULN or 5 x IULN if know liver metastases)
* Otherwise, all acute toxicity at study entry ≤ Grade 1 by NCI CTC v4.0, or recovered to baseline

Exclusion Criteria:

* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men unwilling to use effective contraception during study until conclusion of 12-week post-treatment evaluation period.
* Patients with Gilbert's disease or known CNS metastatic disease. However, patients with CNS metastases who are asymptomatic and have completed a course of therapy are eligible for the study provided that they are clinically stable for 1 month prior to entry as defined as: (1) no evidence of new enlarging CNS metastasis, (2) off steroids or on a stable dose of steroids.
* Patients with CEA plasma levels > 1000 ng/mL must be approved in advance by the Sponsor.
* Patients with active ≥ Grade 3 anorexia, nausea or vomiting, and/or signs of intestinal obstruction.
* Patients with non-melanoma skin cancer or carcinoma in situ of the cervix are eligible, while patients with other prior malignancies must have had at least a 3-year disease-free interval, or are deemed at low risk for recurrence by his/her treating physician.
* Patients known to be HIV positive, hepatitis B positive, or hepatitis C positive.
* Known history of unstable angina, MI, or CHF present within 6 months or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy.
* Known history of clinically significant active COPD, or other moderate-to-severe chronic respiratory illness present within 6 months.
* Infection requiring intravenous antibiotic use within 1 week.
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Safety | Safety will be measured routinely during the 6 months of administration and afterwards during follow-up for up to 5 years
  The primary outcome measured will be safety of IMMU-130 administered at different dose levels. Safety will be assessed by reviewing the number of adverse events and overall toxicity.

SECONDARY OUTCOMES:
Assess PK | Efficacy will be measured every 8 weeks during treatment and every 3 months during the 1st year and then every 6 months up to 5 years thereafter.
  The secondary objectives are to assess pharmacokinetics and immunogenicity, and to obtain preliminary information on efficacy with this dosing schedule. Efficacy will be assessed using CT scan imaging.